CLINICAL TRIAL: NCT00963898
Title: The Clinical Efficacy of the Combination Target Controlled Infusion With Bispectral Index Monitor in Propofol Sedation for Dental Patients With Mental Retardation
Brief Title: Accurate Controlled Dental Sedation
Acronym: ACDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okayama University (Other)
Responsible Party: Department of Dental Anesthesiology, Okayama University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1104mai
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2009-08-24 (Estimated); Status verified 2009-08

CONDITIONS: Mental Retardation
Keywords: Intravenous sedation; Target controlled infusion; Bispectral index; Dental treatment; Mental Retardation; Deep sedation
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mental Retardation (Experimental)
  Interventions: Device: Target controlled infusion(TCI), Bispectral index(BIS)

INTERVENTIONS:
Device: Target controlled infusion(TCI), Bispectral index(BIS) — Using TCI and BIS or not

SUMMARY:
The aim of this study is to evaluate benefits of the method of dental sedation using Target controlled infusion (TCI) combined with Bispectral index (BIS) monitoring in patients with Mental Retardation and challenging behavior.

DETAILED DESCRIPTION:
The intravenous sedation of using of propofol is very effective for dental patients with Mental Retardation and challenging behavior. However, it is very difficult to titrate the dose of propofol for maintaining the adequate sedative depth because of the difficulty of verbal communication with them. Therefore, the infusion of excessive propofol dose elicits the complications and delay of recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 16 or over,
2. American Society of Anesthesiologists (ASA) physical status 1 or 2
3. The treatments of dental caries, endodontics, periodontics and prosthesis were planed
4. Participants had moderate or severe Mental Retardation, and were not completely cooperated with dental treatment

Exclusion Criteria:

1. Patients could communicate and cooperate with dental treatment, but used dental sedation for decrease of the anxiety and the fear about dental treatment or another reasons,
2. Patients needed premedication
3. Patients had uncontrolled or sever medical condition

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The dose of anesthesia agent | 1 day
The recovery times of eyelash reflex and eye opening | 1 day
The time to going home | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Hitoshi Higuchi, D.D.S., Ph.D, Principal Investigator — Okayama University
Locations (1):
- Department of Dental Anesthesiology, Okayama University Hospital, Okayama, Okayama-ken, Japan